CLINICAL TRIAL: NCT05829135
Title: Managing Visual Comfort and Function in Patients With Low Vision Using Acuvue Oasys
Brief Title: Improving Glare and Visual Comfort for Patients With Visual Impairment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: contact lens no longer available for study
Sponsor: Nova Southeastern University (Other)
Collaborators: American Academy of Optometry (Other)
Responsible Party: Principal Investigator, So Yeon Lee, Assistant professor, Nova Southeastern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-128
Record Dates: First submitted 2022-08-25; First posted 2023-04-25 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Photophobia; Visual Impairment; Low Vision
MeSH Terms: conditions — Photophobia; Vision Disorders; Vision, Low

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment group (Experimental): All participants will be fit with Acuvue Oasys with Transitions.
  Interventions: Device: Acuvue Oasys with Transitions

INTERVENTIONS:
Device: Acuvue Oasys with Transitions — soft contact lenses with darkening technology

SUMMARY:
To assess the use of contact lenses with transitions technology to improve glare, light sensitivity and overall visual comfort in patients with visual impairment.

DETAILED DESCRIPTION:
Acuvue Oasys Contact Lenses with Transitions Light Intelligent Technology can adapt to the amount of visible light in the environment, darkening the lenses in bright sunlight, and returning to regular tint in normal or dim environment.

Purpose of this study is to assess whether individuals with visual impairment may benefit from these lenses to minimize glare, light sensitivity symptoms and improve the overall visual comfort.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Able to speak and read English
* Experience glare and light sensitivity that impacts patient's daily living activities
* Have confirmed diagnosis of ocular condition including but not limited to Stargardt's, Cone dystrophy, Cone-rod dystrophy, Albinism, Retinitis Pigmentosa and Achromatopsia.
* Willing and able to wear the contact lenses as instructed

Exclusion Criteria:

* Are pregnant, nursing or planning to become pregnant during the course of the study
* Have current/recent ocular infection, inflammation, surgery in the past 3 months that contraindicates contact lens wear

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Glare test | Measure change from baseline at the 6 week follow-up visit
  Measure visual acuity and contrast sensitivity with or without illumination source

SECONDARY OUTCOMES:
Visual Activities Questionnaire on Glare and Light sensitivity visual functions | Measure change from baseline at the 6 week follow-up visit
  Patient will rate 7 questions on scale ranges from 1-5, higher score indicates more symptoms related to glare and light sensitivity during daily living tasks. Max value 35

CONTACTS AND LOCATIONS:
Overall Officials: So Yeon Lee, OD, Study Chair — Nova Southeastern University
Locations (1):
- Nova Southeastern University, Davie, Florida, United States

IPD SHARING:
Plan to Share IPD: No